CLINICAL TRIAL: NCT02607514
Title: Mechanisms of Hyperthermic Yoga for the Treatment of Depression
Brief Title: Hyperthermic Yoga for Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Maren Nyer, Maren Nyer, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000704; 5K23AT008043-05 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate yoga arm (Experimental): participants will immediately start the 8-week hyperthermic yoga intervention
  Interventions: Behavioral: hyperthermic yoga
- delayed yoga arm (Other): participants will wait 8-weeks to start the 8-week hyperthermic yoga intervention
  Interventions: Behavioral: hyperthermic yoga

INTERVENTIONS:
Behavioral: hyperthermic yoga — heated yoga, 90-minutes
  Other Names: Bikram Yoga

SUMMARY:
Study is a randomized controlled trial to assess the feasibility, acceptability, efficacy, and mechanisms of action of hyperthermic yoga versus a waitlist control for 80 medically healthy adults with mild to moderate depressive symptoms. The primary aim is to test the acceptability and feasibility of hyperthermic yoga as a treatment for depression. The secondary aim is to examine the effect size/efficacy of hyperthermic yoga for depressive symptoms. The tertiary aim is to explore physiological and psychological mechanisms of action.

ELIGIBILITY:
Inclusion Criteria

1. Adults ages 18-60
2. English language proficiency
3. Ability to provide informed consent
4. Score of >23 on the Inventory of Depressive Symptomatology - Clinician Rated (IDS-CR)
5. Able and willing to attend two 90-minute hyperthermic yoga sessions per week
6. Willingness to keep existing exercise regimen (even if that is sedentary) stable over study course
7. Women of childbearing potential must use an acceptable form of birth control
8. Membership to the Bikram Yoga Boston and Bikram Yoga Cambridge studios via studio website "Interested in research" option through a centralized portal (this will remain central until January 1, 2017)
9. Willingness to adhere to hydration requirements (i.e., an additional four 8 oz servings of water pre- and post-yoga classes)

Exclusion Criteria

1. Pregnancy or planned pregnancy during study
2. History of psychiatric hospitalization within the past year
3. Active suicidal intent within the past year ("yes" on item 4 or 5 on the Columbia-Suicide Severity Rating Scale)
4. History of neurologic disorders that could interfere in study participation
5. History of bipolar disorder, psychotic disorders, eating disorders, and/or substance abuse or dependence (within the last year), as per the Mini-International Neuropsychiatric Interview (MINI)
6. Psychotropic medication use that has been stable for <3 months
7. Use of stimulant medications or diet pills during the study, or any pre-workout powders or liquids designed to provide excessive energy
8. Positive urine toxicology screen due to illicit drug use or other exclusionary medications. (Potential false positives will be addressed on a case-by-case basis at the discretion of the investigator)
9. Active conditions which may also cause depressive symptoms (e.g. epilepsy, hypothyroidism)
10. Medical conditions that may make participation unsafe (e.g., diabetes [I & II], cardiovascular disease, hypertension [>140 systolic and/or >90 diastolic], hypotension [<90 systolic and/or <60 diastolic, during screening], orthostatic hypotension [systolic drop of 20 points or 10 point diastolic or heart rate increase by 10], autoimmune disorders, malignancy, or autonomic dysfunction)
11. > 6 one hour classes of meditation or other mind-body disciplines (e.g., Tai chi or yoga) within the last 6 months
12. Current individual or group psychotherapy established for <3 months
13. A subject who in the opinion of the Principal Investigator would not be able to safely complete the study or would jeopardize study integrity
14. History of heat intolerance or heat stroke
15. Unsafe cardiac status as defined by abnormal ECG reading at screening visit as determined by medical monitor, study doctor, or subject's PCP or cardiologist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Depression Clinical and Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nyer MB, Hopkins LB, Nagaswami M, Norton R, Streeter CC, Hoeppner BB, Sorensen CEC, Uebelacker L, Koontz J, Foster S, Dording C, Giollabhui NM, Yeung A, Fisher LB, Cusin C, Jain FA, Pedrelli P, Ding GA, Mason AE, Cassano P, Mehta DH, Sauder C, Raison CL, Miller KK, Fava M, Mischoulon D. A Randomized Controlled Trial of Community-Delivered Heated Hatha Yoga for Moderate-to-Severe Depression. J Clin Psychiatry. 2023 Oct 23;84(6):22m14621. doi: 10.4088/JCP.22m14621. PMID 37883245

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed Yoga Arm: participants will wait 8 weeks to start the 8-week hyperthermic yoga intervention
  hyperthermic yoga: heated yoga, 90-minutes
Period: Overall Study
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Started | 40 | 40
Completed | 22 | 26
Not Completed | 18 | 14

BASELINE CHARACTERISTICS:
Population: The number of baseline participants reported is the sample that we analyzed in our a priori Modified Intent-to-Treat (MITT) primary analysis. A modified intent-to-treat (MITT) approach was used. Analyses only included participants who completed at least one assessment following their initial baseline visit; yoga participants were only included if they completed at least one heated yoga class and subsequent assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11.65) | 33.12 (11.93) | 32.71 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 24 | 21 | 45
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 32 | 65
IDS-CR [Mean (Standard Deviation); unit: units on a scale] — Inventory of Depressive Symptoms - Clinician Rated.
  units on a scale | 36.86 (8.80) | 34.38 (6.68) | 35.63 (7.87)
HAMD-17 [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Scale - 17, range 0-52 (higher is more severe depressive symptoms).
  units on a scale | 22.21 (5.42) | 20.78 (4.02) | 21.51 (4.80)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms as Measured by the Inventory of Depressive Symptomatology - Clinician Rated (IDS-CR)
Description: Inventory of Depressive Symptomatology - Clinician Rated. Scale range: 0-84 (higher = greater depressive symptoms)
Time Frame: 8-week primary endpoint
Population: The number of baseline participants reported is the sample that we analyzed in our a priori Modified Intent-to-Treat (MITT) primary analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 17.93 (12.70) | 29.63 (9.58)

2. Primary Outcome: Feasibility and Tolerability Measured by Percent of the Yoga Group Who Complete a Week 8 Assessment
Description: Measured by percent of the yoga group who complete a week 8 assessment
Time Frame: 8-week primary end point
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
Participants | 27 | 32

3. Primary Outcome: Acceptability as Measured by the Acceptability Interview Completed at 8-week Endpoint or Early Termination
Description: Acceptability Interview: A 19-question qualitative interview assesses perception of ease of participation, program likeability, and perceived benefits of the yoga program. Adapted from DeBoer et al. It was a 1-10 likert scale with 1 = lowest, 10 = highest to rate acceptability of the yoga intervention. These are the items we used: 1) how much did you enjoy the yoga itself?; 2) how much did you enjoy the aftereffects of the yoga?; and 3) how reasonable did you find the time commitment to be?
Time Frame: at the end of 8-weeks or early termination.
Population: we analyzed participants who finished the trial in the immediate yoga arm, delayed yoga arm, or terminated early from the intervention.
  *we only published and analyzed results from the immediate yoga arm
Measure: Mean (Standard Deviation); unit: likert scale units
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 27 | 27
likert scale units
  Enjoyment of yoga | 7.17 (2.28) | 7.52 (1.99)
  Enjoyment of aftereffects of yoga | 8.33 (1.74) | 8.59 (1.67)
  Reasonable time commitment | 6.90 (2.38) | 7 (2)

4. Secondary Outcome: Quality of Life as Measured by the Quality of Life Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) Over 8 Weeks.
Description: Quality of Life Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) Range 0-70 with higher scores indicating greater life satisfaction and enjoyment
Time Frame: 8-weeks end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 51.33 (7.90) | 41.34 (8.24)

5. Secondary Outcome: General Health as Measured by the Medical Outcomes Study 36-item Short-form Survey (SF-36)
Description: Medical Outcomes Study 36-item short-form survey (SF-36): Assesses bodily pain, general health perception, vitality, social functioning, physical and emotional impediments to role functioning, mental health, and includes an overall physical component scale (PCS) and mental component scale (MCS).
  scores range from 0-100 with 100 being the best.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 61.67 (23.15) | 53.5 (18.72)

6. Secondary Outcome: Physical Functioning as Measured by the Physical Component Scale (PCS) of the Medical Outcomes Study 36-item Short-form Survey (SF-36) Over 8 Weeks.
Description: Medical Outcomes Study 36-item short-form survey (SF-36)86: Assesses bodily pain, general health perception, vitality, social functioning, physical and emotional impediments to role functioning, mental health, and includes an overall physical component scale (PCS) and mental component scale (MCS).
  Scores range from 0-100 with 100 being the best.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 47.62 (10) | 53.33 (16)

7. Secondary Outcome: Perceived Stress as Measured by the Perceived Stress Scale (PSS) Over 8 Weeks.
Description: The Perceived Stress Scale (PSS): Measures perceived level of stress. Scale range: 0-40 (higher = more perceived stress)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 17.42 (8.22) | 22.33 (5.84)

8. Secondary Outcome: Anxiety as Measured by the Spielberger State-Trait Anxiety Inventory (STAI), State, Over 8 Weeks.
Description: Spielberger State-Trait Anxiety Inventory (STAI), State. A 40-item commonly used measure that distinguishes between state vs. trait anxiety.
  Ranges from 0-63 with higher scores indicating more anxiety.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 40.69 (10.74) | 48.43 (9.66)

9. Secondary Outcome: Sleep as Measured by the Pittsburg Sleep Quality Index (PSQI): A Commonly Used and Well-validated Self-rated Measure of Sleep-quality and Disturbance Over 8-weeks.
Description: Pittsburg Sleep Quality Index (PSQI): A commonly used and well-validated self-rated measure of sleep-quality and disturbance.
  total score ranges from 0-21 with higher score indicating worse sleep quality.
Time Frame: 8-weeks
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Long Term Effects of Heated Yoga Intervention as Measured by All Primary and Secondary Outcomes After 1 Month Post-intervention.
Description: see all primary and secondary outcome measures listed here.
Time Frame: one month post intervention
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Anxiety as Measured by the Spielberger State-Trait Anxiety Inventory (STAI), Trait, Over 8 Weeks.
Description: Spielberger State-Trait Anxiety Inventory (STAI), Trait. A 40-item commonly used measure that distinguishes between state vs. trait anxiety.
  Ranges from 0-63 with higher scores indicating more anxiety.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 46.70 (11.80) | 54.1 (8.25)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Immediate Yoga Arm | Delayed Yoga Arm
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 3/33 | 1/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Yoga Arm (N=33) | Delayed Yoga Arm (N=32)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT02607514/Prot_SAP_000.pdf